CLINICAL TRIAL: NCT06442904
Title: A Digital Education Program in Oral and Maxillofacial Radiology: Effect on Image Quality Evaluated in a Cluster Randomized Controlled Trial
Brief Title: Can a Digital Education Program in Radiographic Imaging Technique for Dental Professionals Improve Image Quality?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Västerbotten County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Maria Garoff, Associate professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Umea University, Sweden
Record Dates: First submitted 2024-05-30; First posted 2024-06-04 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Radiography; Dentistry
Keywords: digital education; oral and maxillofacial radiology

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Access to a digital education program for three months.
  Interventions: Other: Digital education program
- Control group (No Intervention): The control group is not offered any intervention.

INTERVENTIONS:
Other: Digital education program — The approximately six hours long digital education program will be available for three months and implies further education in intraoral radiographic examinations.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn if a digital education program designed for dental professionals can lead to radiographic examinations of better quality. The main questions it aims to answer are:

Does the digital education program lead to more radiographic examinations of good quality? Does the digital education program lead to better theoretical and practical understanding regarding image quality among dental professionals?

Researchers will compare answers from a theoretical test and image quality in radiographic examinations between participants with respectively without access to the digital education program.

Participants will:

* have access to the digital education program for three months
* after three months all study participants are invited to answer a theoretical test

DETAILED DESCRIPTION:
The present study aims to evaluate a digital education programs effect on image quality in intraoral radiographic examinations performed by dental professionals. The present study is part of an on-going cross sectional descriptive project where dental professionals employed in general dental care in the county of Västerbotten, Sweden constitute the study population. The purpose of the project is to gain a broader understanding of a digital education programs impact on the theoretical and practical competencies among dental professionals regarding intraoral dental radiographic examinations.

Approximately 80 dental professionals have provided written informed consent regarding study participation. In the present study, approximately 40 participants will for three months be offered the intervention and join a digital education program. Approximately 40 participants will during the same period not be offered the intervention and constitute the control group. Effects on practical competencies between groups will be evaluated when analyzing image quality of intraoral radiographic examinations. Effects on theoretical competencies between groups will be analyzed with a theoretical test.

Cluster randomization of dental clinics will be made for study included participants to either intervention group or control group. Recruitment of study participants will end in August 2024.

The investigators hypothesize that the digital education program will improve the theoretical competence and radiographic image quality in intraoral radiographic examinations.

ELIGIBILITY:
Inclusion Criteria:

• Dental professionals performing radiographic examinations employed in general dentistry in the County Council of Västerbotten, Sweden

Exclusion Criteria:

• Dental professionals not performing radiographic examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Image quality | Baseline and three months post-intervention
  Change in image quality of intraoral radiographic examinations measured with a protocol designed for diagnostic image quality assessment. Comparisons between intervention- and control group will be made.

SECONDARY OUTCOMES:
Theoretical competence | One month post-intervention
  Change in theoretical competence measured in a theoretical test. Comparisons between intervention- and control group will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Garoff, Assoc. Prof., Principal Investigator — Umeå University
Locations (1):
- Folktandvården Region Västerbotten, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No